CLINICAL TRIAL: NCT02241070
Title: The Potential for Mindfulness-Based Intervention in Workplace Mental Health Promotion: Results of a Randomized Controlled Trial
Brief Title: The Potential for Mindfulness-Based Intervention in Workplace Mental Health Promotion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Collaborators: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, GCRC, Chung Shan Medical University, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCH 110606
Record Dates: First submitted 2014-09-07; First posted 2014-09-16 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Mental Health Wellness 1
Keywords: mindfulness meditation; mental health promotion; worker

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mindulness-based intervention (Experimental): Mindulness-based intervention was eight weeks of mindfulness training with forty-five minutes of homework practice every day during the training course. A leader and a professional facilitator led the group. The leader was a long-term mindfulness and vipassana meditation trainer who had practiced both types of meditation for more than two decades and had completed mindfulness trainer education; the professional facilitator was a mindfulness practitioner and a psychiatrist. The group met weekly for two hours in-session at the workplace.
  Interventions: Behavioral: mindulness-based intervention
- waiting-list control (No Intervention): passive control group

INTERVENTIONS:
Behavioral: mindulness-based intervention — A number of mindfulness techniques, including both "formal" and "informal" practices with integration in the context of Mind/Body meditation, were explored in order to cultivate moment-by-moment present awareness with non-judgmental acceptance.
  Arms: mindulness-based intervention

SUMMARY:
The aims of the study are to determine the effectiveness of Mindfulness-Based Interventionas a workplace health promotion program on psychological distress, prolonged fatigue, job strain (job control and job demand), and perceived stress and to explore the influences of personal characteristics (including gender, age, education, and occupation) on the outcomes of the intervention with time.

DETAILED DESCRIPTION:
This study was one component of the Taiwan Workplace Mental Health Promotion Scheme. The study adopted a study design of a randomized controlled trial. Two large-scale manufacturing factories were chosen for this study. All of the factories' 3270 full-time employees were requested to fill in a questionnaire comprising questions regarding mental health and job strain. Of these employees, 2849 individuals were willing to complete the questionnaire. A total of 431 employees (15.13%) were found to be in psychological distress with job strain. The screening procedure was carried out between June and July in 2011. A letter of invitation with an introduction to MBI was sent to these employees. Of these 431 employees, only 144 responded that they would be willing to take part voluntarily in the study. These 144 workers were allocated randomly into the intervention group (Group I, n=72) or the waiting-list control group (Group C, n=72).

All the participants were measured five times with an interval of four weeks between measurements. These measurements were taken at pre-intervention (T1), at mid-intervention (T2), at the completion of intervention (T3), four weeks after intervention (T4), and eight weeks after intervention (T5). The data related with the effectiveness of the intervention were obtained between August and December in 2011.

ELIGIBILITY:
Inclusion Criteria:

* Healthy employees with psychological distress and job strain
* Full-time paid workers

Exclusion Criteria:

* Age < 18y or > 65y
* Part-time workers
* The workers are not willing to take part in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
psychological distress | four months
  Psychological distress was measured by the Chinese Health Questionnaire (CHQ-12), a well-validated instrument

SECONDARY OUTCOMES:
prolonged fatigue | Four months
  Prolonged fatigue was measured by The Checklist Individual Strength questionnaire (CIS), which confirmed discriminant validity and convergent validity.
job strain | four months
  The Job Content Questionnaire (JCQ) was used to assess job control and job demands (job strain).
perceived stress | four months
  The 10-item Perceived Stress Scale (PSS-10) was adopted to measure a global level of perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Cheng Tang, MD; PhD, Principal Investigator — Changhua Christian Hospital
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan

REFERENCES:
- [Derived] Huang SL, Li RH, Huang FY, Tang FC. The Potential for Mindfulness-Based Intervention in Workplace Mental Health Promotion: Results of a Randomized Controlled Trial. PLoS One. 2015 Sep 14;10(9):e0138089. doi: 10.1371/journal.pone.0138089. eCollection 2015. PMID 26367270